CLINICAL TRIAL: NCT04951648
Title: A Randomized Controlled, Open-lable, Phase III, Multicenter Clinical Study of Almonertinib Versus Platinum-based Chemotherapy as First-line Therapy in Patients With Locally Advanced or Metastatic NSCLC Harbouring Uncommon EGFR Mutation
Brief Title: A Phase III Study to Assess the Efficacy and Safety of Almonertinib Versus Platinum-based Chemotherapy as First-line Therapy in Patients With Locally Advanced or Metastatic NSCLC Harbouring Uncommon EGFR Mutation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10296-305
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Phase III, NSCLC, Almonertinib, uncommon EGFR mutation, first-line therapy，platinum-based chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonertinib (Experimental)
  Interventions: Drug: Almonertinib
- Platinum-based doublet chemotherapy (Active Comparator)
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: Almonertinib — Almonertinib 165 mg，orally once a day Treatment can continue until disease progression, unacceptable toxicity or other discontinuation criteria are met.
  Other Names: HS-10296
  Arms: Almonertinib
Drug: chemotherapy — Pemetrexed (500mg/m2) plus Carboplatin (AUC5)or Pemetrexed (500mg/m2) plus Cisplatin (75mg/m2) on Day 1 of 21day cycles (every 3 weeks) for 4~6 cycles, followed by pemetrexed mainten-ance therapy every 3 weeks until disease progress-ssion, unacceptable toxicity or other discontinuation criteria are met.
  Arms: Platinum-based doublet chemotherapy

SUMMARY:
To assess the efficacy and safety of Almonertinib versus platinum-based chemotherapy as first-line therapy in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring uncommon EGFR mutation.

DETAILED DESCRIPTION:
This is a randomized, open-lable, multicenter, phase III study to assess the efficacy and safety of Almonertinib versus platinum-based chemotherapy as first-line therapy in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring at least one uncommon EGFR mutation, including L861Q, G719X or S768I. Patients who have not received any systemic treatment to receive Almonertinib or platinum-based chemotherapy in a 1:1 ratio, and treatment will be continued until disease progression, unacceptable toxicity or other discontinuation criteria are met. After progression, patients may receive Almonertinib for as long as their treating physician considers they are deriving clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are willing to participate in this clinical study, understand the study procedures and are able to sign the informed consent in person.
2. Age at least 18 years.
3. Histologically or cytologically confirmed diagnosis of primary non-small lung cancer (NSCLC), histologically confirmed non-squamous pathology.
4. Locally advanced or metastatic NSCLC.
5. Patients must be treatment-naïve for locally advanced or metastatic NSCLC.
6. The tumor harbors uncommon EGFR mutations (one of the following EGFR mutation: L861Q, G719X or S768I), assessed by Xiamen AmoyDx EGFR (ADx-ARMS, Super-ARMS method) kit in central laboratory.
7. Measurable disease by RECIST 1.1.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Female patients should be using adequate contraceptive measures and should not be breastfeeding during the study and six months after the last dosing of study. Male patients should be willing to use barrier contraception (condoms) during the study and six months after the last dosing of study.
10. A pregnancy test should be done before randomization unless having an evidence of non-child-bearing potential.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Prior treatment with EGFR-TKI therapy.
   2. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks prior to randomization.
   3. The presence of pleural effusion/peritoneal effusion/pericardial effusion requiring clinical intervention.
   4. Major surgery within 4 weeks prior to randomization.
   5. Spinal cord compression or unstable brain metastasis; Meningeal or brainstem metastases.
   6. Patients had received medications or herbal supplements known to be strong inducers and inhibitors of cytochrome CYP3A4 within 7 days prior to randomization or required to continue these agents during the study period.
   7. Patients are receiving medications known to prolong QT interval or may cause tip torsion ventricular tachycardia, or are still in the washout period (relatively random phase), or need to be continued during the study period.
   8. Patients were subjects in another clinical trial within 4 weeks prior to randomization or patients were within 5 half-lives of any other investigational agent.
2. Any unresolved toxicity Common Terminology Criteria for Adverse Events (CTCAE) ≥ Grade 2 from the prior anticancer therapy.
3. Inadequate bone marrow reserve or organ function.
4. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., PR interval > 250 ms).
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure or any concomitant medication known to prolong the QT interval.
   4. Left ventricular ejection fraction (LVEF) <50%.
5. History of other malignancies, excluding fully treated non-melanoma skin cancer, Malignant freckled nevus, in-situ cancer, other solid tumors that hadn't been recurrent for > 5 years following the end of treatment, or local prostate cancer after radical resection.
6. Any evidence of severe or uncontrolled systemic diseases (including uncontrolled hypertension and active bleeding diatheses) or active infection (including hepatitis B, hepatitis C, and human immunodeficiency virus (HIV), etc.).
7. Acquired or congenital immune deficiency diseases, or history of organ transplantation.
8. Serious gastrointestinal function abnormalities that may interfere with drug ingestion, transport, or absorption.
9. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
10. Pregnant or lactating, or intending to become pregnant during the study
11. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
12. Any disease or condition that, in the opinion of the investigator, would compromise the safety of the patient or interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2023-10-04 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by IRC (Independent Review Committee) | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  PFS is defined as the time from randomization until the date of objective disease progression or death regardless of whether the patient withdraws from randomised therapy or receives another anti-cancer therapy prior to progression, based on blinded independent central review assessment according to RECIST 1.1.

SECONDARY OUTCOMES:
PFS assessed by INVs (Investigators) | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  PFS is defined as the time from randomization until the date of disease progression as assessed by INVs according to RECIST 1.1 or death from any cause on study.
Objective response rate (ORR) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  ORR is defined as the number (%) of patients with at least 1 visit response of CR (Complete response) or PR (Partial response) based on blinded independent central review assessment according to RECIST 1.1.
Duration of response (DoR) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  DoR is defined as the time from date for first documented response of until the documented response of progression per RECIST 1.1 or death in the absence of progression based on blinded independent central review assessment.
Disease control rate (DCR) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 2 years.
  DCR is defined as the percentage of patients who have a best overall response of CR or PR or SD based on blinded independent central review assessment according to RECIST 1.1.
Depth of response (DepOR) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression; up to a maximum of approximately 3 years.
  DepOR is defined as the change amount of the sum of the lengths of the longest diameters of the target lesions on blinded independent central review assessment according to RECIST 1.1 in the absence of New Lesions (NLs) or progression of Non-Target Lesions when compared to baseline.
Proportion of patients alive and progression free at 6 months (APF6) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed until 6 months post-randomization.
  APF6 is defined as the percentage (%) of patients who were alive and progression free per RECIST 1.1 at 6 months after randomization.
Proportion of patients alive and progression free at 9 months (APF9) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed until 9 months post-randomization.
  APF9 is defined as the percentage (%) of patients who were alive and progression free per RECIST 1.1 at 9 months after randomization.
Proportion of patients alive and progression free at 12 months (APF12) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed until 12 months post-randomization.
  APF12 is defined as the percentage (%) of patients who were alive and progression free per RECIST 1.1 at 12 months after randomization.
Proportion of patients alive and progression free at 24 months (APF24) assessed by IRC | Tumor scans performed at baseline then every ~6 weeks up to 48 weeks, then every ~12 weeks thereafter until confirmed disease progression. Assessed until 24 months post-randomization.
  APF24 is defined as the percentage (%) of patients who were alive and progression free per RECIST 1.1 at 24 months after randomization.
Overall survival (OS) | From the date of randomization until death due to any cause; up to a maximum of approximately 3 years.
  OS is deﬁned as the time from the date of randomization until death due to any cause.
Percentage of patients alive at 36 months (OS36) | From randomization until death due to any cause, up to a maximum of approximately 3 years.
  OS36 was defined as the percentage (%) of patients who were alive at 36 months after randomization per the Kaplan-Meier estimate of OS at 36 months.
Incidence of Adverse Events (AEs) | From the screening period to 28 days after treatment completion, approximately 3 years.
  AEs are graded according to CTCAE v5.0 and recorded in the case report form.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen Univerisity Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided